CLINICAL TRIAL: NCT01173939
Title: Primary Prevention of MACE With Standard and Intensive Statin Treatment in Hypercholesterolemia Patients With Concomitant Diabetes and Hypertension
Brief Title: Primary Prevention of Major Adverse Cardiac Events (MACE) With Standard and Intensive Statin Treatment in Patients With Diabetes: Survival and Cardiovascular Event Assessments
Acronym: POSITIVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: With recommendation from IDMC, Steering Committee terminated this trial due to ethical concerns raised by J-ART study.
Sponsor: Positive Trial Group (Other)
Responsible Party: Hisao Ogawa, Department of Cardiovascular Medicine, Faculty of Graduate School of Medical Sciences, Kumamoto University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0035
Record Dates: First submitted 2010-07-27; First posted 2010-08-02 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2010-11

CONDITIONS: Hypercholesterolemia; Type 2 Diabetes; Hypertension
Keywords: Hypercholesterolemia with concomitant type 2 diabetes and hypertension
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus, Type 2; Hypertension | interventions — Pravastatin; Rosuvastatin Calcium

ARMS (2):
- Active comparator: Standard Pravastatin Group (Active Comparator)
  Interventions: Drug: Pravastatin
- Intensive Rosuvastatin Group (Active Comparator)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Pravastatin — 5 mg/day or 10 mg/day of pravastatin will be administered orally for 36 months, with a follow-up period of one month. If the target LDL-C level is not attained after one month of treatment, the steps will be taken to reduce the LDL-C to the target level of <120 mg/dL (JASGL 2007 target level) as quickly as possible. (Maximum dose increase of pravastatin: 20 mg/day)
  Arms: Active comparator: Standard Pravastatin Group
Drug: Rosuvastatin — 5 mg/day or 10 mg/day of rosuvastatin will be administered orally for 36 months based on the LDL-C level of the subject, with a follow-up period of one month. If the target LDL-C level is not attained after one month of treatment, the steps will be taken to reduce the LDL-C to the target level of <70 mg/dL as quickly as possible. (Maximum dose increase to rosuvastatin: 20 mg/day)
  Arms: Intensive Rosuvastatin Group

SUMMARY:
The study is being conducted to compare the effect of standard treatment (target LDL-C level: <120 mg/dL (JASGL 2007 target level)) and intensive treatment (target LDL-C level: <70 mg/dL) in the prevention of major adverse cardiac events (MACE) in hypercholesterolemia patients with concomitant type 2 diabetes and hypertension.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following inclusion criteria will be included in the study:

1. Patients giving voluntary written consent to participate in the study
2. Male or female patients 50 years of age or older (at informed consent)
3. Hypercholesterolemia patients (Untreated patients: LDL-C level ≥140 mg/dL; treated patients: LDL-C level ≥120 mg/dL)
4. Type 2 diabetes patients (HbA1c level ≥6.1% (JDS criteria), with or without history of drug therapy)
5. Hypertension patients (SBP ≥130 mmHg or DBP ≥80 mmHg, with or without history of drug therapy)
6. Patients with two or more of the following risk factors

   * Male
   * 65 years of age or older
   * Smoker
   * L/H ratio: ≥3.0 •HbA1c level: ≥8.0%
   * Left ventricular hypertrophy
   * First- or second-degree family history of MACE
   * Microalbuminuria (quantitative testing: ≥30 mg/dL), proteinuria (qualitative testing: + or higher) or eGFR (<60 mL/min/1.73 m2)

Exclusion Criteria:

Patients meeting the following criteria will be excluded from the study:

1. Patients receiving rosuvastatin, pitavastatin, or atorvastatin therapy within one month prior to informed consent
2. Patients judged to have familial hypercholesterolemia
3. Patients with a serum triglyceride level of ≥400 mg/dL
4. Patients with a history of myocardial infarction
5. Patients with a history of coronary revascularization (PCI or CABG)
6. Patients with a history of treatment of unstable angina
7. Patients with a history of cerebrovascular accident (excluding asymptomatic lacunar infarction)
8. Heart failure patients
9. Patients with a history of hypersensitivity to statins
10. Patients with a history of drug-induced myopathy
11. Patients with poorly controlled arrhythmia
12. Patients with severe liver or kidney disease
13. Patients with serious concurrent disease, such as malignancy, or patients with severely limited lifespan
14. Patients who are or may be pregnant
15. Patients judged by the investigators to be ineligible for participation in the study for any other reason

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | At baseline
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | 1 month after treatment initiation
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | 3 month after treatment initiation
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | 6 month after treatment initiation
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | 12 month after treatment initiation
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | 36 month after treatment initiation
MACE (time to event): MACE (time to event): myocardial infarction, unstable angina, cardiovascular death, revascularization, fatal/nonfatal cerebrovascular accident, peripheral arteriopathy, aortic event | At the end of the study or discontinuation up to 4 years

SECONDARY OUTCOMES:
Prevention of individual MACE | At baseline
Prevention of MACE(combination of each category) | At baseline
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | At baseline
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | At baseline
Frequency and distribution of type of deaths during the study period | At baseline
Frequency and distribution of type of hospitalizations during the study period | At baseline
Frequency of other events (malignancy, dementia, need of nursing care) | At baseline
Frequency and type of adverse events | At baseline
Prevention of individual MACE | 1 month after treatment initiation
Prevention of individual MACE | 3 month after treatment initiation
Prevention of individual MACE | 6 month after treatment initiation
Prevention of individual MACE | 12 month after treatment initiation
Prevention of individual MACE | 36 month after treatment initiation
Prevention of individual MACE | At the end of the study (or discontinuation)
Prevention of MACE(combination of each category) | 1 month after treatment initiation
Prevention of MACE(combination of each category) | 3 month after treatment initiation
Prevention of MACE(combination of each category) | 6 month after treatment initiation
Prevention of MACE(combination of each category) | 12 month after treatment initiation
Prevention of MACE(combination of each category) | 36 month after treatment initiation
Prevention of MACE(combination of each category) | At the end of the study (or discontinuation)
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | 1 month after treatment initiation
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | 3 month after treatment initiation
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | 6 month after treatment initiation
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | 12 month after treatment initiation
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | 36 month after treatment initiation
Prevention, frequency and distribution of type of the following non-MACE cardiac and cerebrovascular events during the study period: heart failure requiring hospitalization, transient ischemic attack (TIA), abnormal ankle-brachial index (abnormal ABI) | At study completion up to 4 years
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | 1 month after treatment initiation
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | 3 month after treatment initiation
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | 6 month after treatment initiation
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | 12 month after treatment initiation
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | 36 month after treatment initiation
Frequency and distribution of type of MACE during the study period Including correlation with LDL-C, HDL-C and LDL-C/HDL-C ratio (hereafter referred to as "L/H ratio") | At the end of the study or discontinuation up to 4 years
Frequency and distribution of type of deaths during the study period | 1 month after treatment initiation
Frequency and distribution of type of deaths during the study period | 3 month after treatment initiation
Frequency and distribution of type of deaths during the study period | 6 month after treatment initiation
Frequency and distribution of type of deaths during the study period | 12 month after treatment initiation
Frequency and distribution of type of deaths during the study period | 36 month after treatment initiation
Frequency and distribution of type of deaths during the study period | At the end of the study or discontinuation up to 4 years
Frequency and distribution of type of hospitalizations during the study period | 1 month after treatment initiation
Frequency and distribution of type of hospitalizations during the study period | 3 month after treatment initiation
Frequency and distribution of type of hospitalizations during the study period | 6 month after treatment initiation
Frequency and distribution of type of hospitalizations during the study period | 12 month after treatment initiation
Frequency and distribution of type of hospitalizations during the study period | 36 month after treatment initiation
Frequency and distribution of type of hospitalizations during the study period | At the end of the study or discontinuation up to 4 years
Frequency of other events (malignancy, dementia, need of nursing care) | 1 month after treatment initiation
Frequency of other events (malignancy, dementia, need of nursing care) | 3 month after treatment initiation
Frequency of other events (malignancy, dementia, need of nursing care) | 6 month after treatment initiation
Frequency of other events (malignancy, dementia, need of nursing care) | 12 month after treatment initiation
Frequency of other events (malignancy, dementia, need of nursing care) | 36 month after treatment initiation
Frequency of other events (malignancy, dementia, need of nursing care) | At the end of the study or discontinuation up to 4 years
Frequency and type of adverse events | 1 month after treatment initiation
Frequency and type of adverse events | 3 month after treatment initiation
Frequency and type of adverse events | 6 month after treatment initiation
Frequency and type of adverse events | 12 month after treatment initiation
Frequency and type of adverse events | 36 month after treatment initiation
Frequency and type of adverse events | At the end of the study or discontinuation up to 4 years

CONTACTS AND LOCATIONS:
Locations (317):
- Japan (317):
  - Hiramitsu Heart Clinic, Nagoya, Aichi Pref.
  - Medical Dock&Clinic, Nagoya, Aichi Pref.
  - Matsuno Medical Clinic, Iyo Gun, Ehime Pref.
  - Ishite Matsumoto Naika Junkanki Clinic, Matsuyama, Ehime Pref.
  - Ehime Medical CO-OP Izumigawa Clinic, Niihama, Ehime Pref.
  - Tsugawa Internal Medicine Clinic, Echizen, Fukui Pref.
  - Fukui Chuo Clinic, Fukui, Fukui Pref.
  - Koshino Clinic, Sakai, Fukui Pref.
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka Pref.
  - Saiseikai Futsukaichi Hospital, Chikushino-shi, Fukuoka Pref.
  - Abies Clinic, Fukuoka, Fukuoka Pref.
  - Hirano Medical Clinic, Fukuoka, Fukuoka Pref.
  - Naitoh Clinic, Fukuoka, Fukuoka Pref.
  - Saku Hospital, Fukuoka, Fukuoka Pref.
  - Fukuoka Tokushukai Medical Center, Kasuga, Fukuoka Pref.
  - Morizono Naika, Kitakyushu, Fukuoka Pref.
  - Kawai Naika Clinic, Gifu, Gifu Pref.
  - Hiroshima General Hospital of West Japan Railway Company, Hiroshima, Hiroshima Pref.
  - Hijirigaoka Hospital, Date, Hokkaido Pref.
  - Kyoaikai Hospital, Hakodate, Hokkaido Pref.
  - Miyazawa Cardiovascular And Internal Medicine Clinic, Kato-gun, Hokkaido Pref.
  - Jiyugaoka Yamada Clinic, Obihiro, Hokkaido Pref.
  - Chikama Clinic, Sapporo, Hokkaido Pref.
  - Hiro Clinic, Sapporo, Hokkaido Pref.
  - Medical and Radiology Clinic Caress Sapporo Hokko Memorial Hospital, Sapporo, Hokkaido Pref.
  - Seiwa Memorial Hospital, Sapporo, Hokkaido Pref.
  - Medical Treatment Corporate Foundation Yubari Kibounomori Yubari City Clinic, Yūbari, Hokkaido Pref.
  - Ino Hospital, Himeji, Hyogo Pref.
  - Katsuya Clinic, Amagasaki, Hyogo Pref
  - Kotani Diabetes Clinic, Kobe, Hyogo Pref
  - Shimizu Clinic, Kobe, Hyogo Pref
  - Dr. Kodama's Office of Internal Medicine, Nishinomiya, Hyogo Pref
  - Koga Hospital, Koga, Ibaraki Pref.
  - Imura Internal Medicine Clinic, Hakusan, Ishikawa Pref.
  - Yanagi Medical Clinic, Hakusan, Ishikawa Pref.
  - Okyozuka Clinic, Ishikawa Gun, Ishikawa Pref.
  - Koni Clinic, Kahoku Gun, Ishikawa Pref.
  - Murata Clinic, Kahoku Gun, Ishikawa Pref.
  - Arai Naika Clinic, Kanazawa, Ishikawa Pref.
  - Dr. Hayakawa's Family Clinic, Kanazawa, Ishikawa Pref.
  - Wakasa Medical Clinic, Kanazawa, Ishikawa Pref.
  - Morita Hospital, Komatsu, Ishikawa Pref.
  - Kawasaki Family Clinic, Ichinoseki, Iwate Pref.
  - Sugie Clinic, Iwate Gun, Iwate Pref.
  - Katsura General Clinic, Morioka, Iwate Pref.
  - Takamiya General Clinic, Shiwa Gun, Iwate Pref.
  - Hayashi Clinic, Marugame, Kagawa Pref.
  - Otsuka Internal Medicine Clinic, Marugame, Kagawa Pref.
  - Center for Preventive Medical Treatment, NTT West Takamatsu Hospital, Takamatsu, Kagawa Pref.
  - Hananomiya Clinic, Takamatsu, Kagawa Pref.
  - Hasegawa Outpatients Clinic for Cardiovascular Disease, Takamatsu, Kagawa Pref.
  - Kojima Clinic, Takamatsu, Kagawa Pref.
  - Matsuoka Clinic, Takamatsu, Kagawa Pref.
  - Osumi-Kanoya Hospital, Kanoya, Kagoshima Pref.
  - Yakushima Tokushukai Hospital, Kumage Gun, Kagoshima Pref.
  - Nemoto G.I.M. Clinic, Ashigara-kami Gun, Kanagawa Pref.
  - Magokoro Internal Medicine and Orthopedic Clinic, Ashigarakami Gun, Kanagawa Pref.
  - Kasuya Clinic, Atsugi, Kanagawa Pref.
  - Kuboshima Clinic, Fujisawa, Kanagawa Pref.
  - Takahashi Clinic, Fujisawa, Kanagawa Pref.
  - Akizawa Clinic, Isehara, Kanagawa Pref.
  - Medical Corp Takeda Clinic, Isehara, Kanagawa Pref.
  - Hashimoto Clinic, Kamakura, Kanagawa Pref.
  - Iroden Clinic, Kamakura, Kanagawa Pref.
  - Kamakura Naika Shinryosyo, Kamakura, Kanagawa Pref.
  - Shohei Clinic, Kamakura, Kanagawa Pref.
  - Hatori Medical Clinic, Kawasaki, Kanagawa Pref.
  - Hirayasu Iin, Kawasaki, Kanagawa Pref.
  - Kamegaya Medical Clinic, Kawasaki, Kanagawa Pref.
  - Kirimura Iin, Kawasaki, Kanagawa Pref.
  - Kojima Clinic, Odawara, Kanagawa Pref.
  - Hakuai Iin, Sagamihara, Kanagawa Pref.
  - Sato Clinic, Sagamihara, Kanagawa Pref.
  - Toshiba Rinkan Hospital, Sagamihara, Kanagawa Pref.
  - Yamamoto Clinic, Sagamihara, Kanagawa Pref.
  - Fukumura Clinic, Yokohama, Kanagawa Pref.
  - Fukushi Clinic, Yokohama, Kanagawa Pref.
  - International Goodwill Hospital, Yokohama, Kanagawa Pref.
  - Kikuchi Clinic, Yokohama, Kanagawa Pref.
  - Matsuo Naika Clinic, Yokohama, Kanagawa Pref.
  - Miho-cho Cardiovascular Medical Clinic, Yokohama, Kanagawa Pref.
  - Minamisawa Clinic, Yokohama, Kanagawa Pref.
  - Miyoshi-Clinic, Yokohama, Kanagawa Pref.
  - Paula's Clinic, Yokohama, Kanagawa Pref.
  - Shimokurata Heart Clinic, Yokohama, Kanagawa Pref.
  - Shinwakai Fukuda Iin, Yokohama, Kanagawa Pref.
  - Shinyoshida Clinic, Yokohama, Kanagawa Pref.
  - Suzuki Orthopedic Clinic, Yokohama, Kanagawa Pref.
  - Yokohama City University Medical Center, Yokohama, Kanagawa Pref.
  - Yokohama Sotetsu bldg. clinic of internal medicine, Yokohama, Kanagawa Pref.
  - Hara Clinic, Yokosuka, Kanagawa Pref.
  - Ueta Medical Clinic, Kochi, Kochi Pref.
  - Nakayama Cardiovascular Clinic, Amakusa, Kumamoto Pref.
  - Yamashita Clinic, Amakusa, Kumamoto Pref.
  - National Health Insurance Central Hospital Aso, Aso, Kumamoto Pref.
  - Sakanashi Heart Clinic, Aso, Kumamoto Pref.
  - Koyasako iin, Kamimashiki Gun, Kumamoto Pref.
  - Kawaguchi Hospital, Kikuchi, Kumamoto Pref.
  - Miyamoto Internal Clinic, Kikuchi, Kumamoto Pref.
  - Doi Cardiovascular Clinic, Kumamoto, Kumamoto Pref.
  - Doi Naika-ichoka Clinic, Kumamoto, Kumamoto Pref.
  - Haraguchi Circular&Internal Medical Clinic, Kumamoto, Kumamoto Pref.
  - Jinnouchi Clinic Diabetes Care Center, Kumamoto, Kumamoto Pref.
  - Kiyota Junkanki Naika Iin, Kumamoto, Kumamoto Pref.
  - Maki Cardiovascular Clinic, Kumamoto, Kumamoto Pref.
  - Nozuhara Clinic, Kumamoto, Kumamoto Pref.
  - Ootsuka Hospital, Kumamoto, Kumamoto Pref.
  - Shono Heart Clinic, Kumamoto, Kumamoto Pref.
  - Suefuji Naika Junkankika, Kumamoto, Kumamoto Pref.
  - Suizenji Tohya Hospital, Kumamoto, Kumamoto Pref.
  - Terao Hospital, Kumamoto, Kumamoto Pref.
  - Yi Medical Clinic, Kumamoto, Kumamoto Pref.
  - Munakata Clinic, Shimomashiki Gun, Kumamoto Pref.
  - Higashi Diabetes and Cardiovascular Clinic, Tamana, Kumamoto Pref.
  - Yoshimura Jyunnkannkika Naika Iinn, Tamana, Kumamoto Pref.
  - Universal Shipbuilding Co. Ariake Shipyard Ariake Infirmary, Tamana Gun, Kumamoto Pref.
  - Miyagi Clinic Cardiovascular Medicine, Yatsushiro, Kumamoto Pref.
  - Koide Iin, Kizugawa, Kyoto Pref.
  - Asamoto Clinic of Internal Medicine, Kyoto, Kyoto Pref.
  - Gotoh Clinic, Kyoto, Kyoto Pref.
  - Higashiyama Takeda Hospital, Kyoto, Kyoto Pref.
  - Isoda Internal Medical Clinic, Kyoto, Kyoto Pref.
  - Omoto Clinic, Kyoto, Kyoto Pref.
  - Sakazaki Clinic, Kyoto, Kyoto Pref.
  - Shinya Clinic, Kyoto, Kyoto Pref.
  - Takagi Cardiology Clinic, Kyoto, Kyoto Pref.
  - Takenaka Clinic, Kyoto, Kyoto Pref.
  - Tegoshi Clinic, Kyoto, Kyoto Pref.
  - Sawai medical Clinic, Kyōtanabe, Kyoto Pref.
  - Kimura Naika Clinic, Yosa Gun, Kyoto Pref.
  - Shimizu Clinic, Ise, Mie Pref.
  - Horii Clinic Kiodai, Nabari, Mie Pref.
  - Yamoto-naika Clinic, Higashi Matsushima City, Miyagi Pref.
  - Seisuikai Yoshioka QQ Clinic, Kurokawa Gun, Miyagi Pref.
  - Ohtomo Clinic, Tome, Miyagi Pref.
  - Shimoina Kosei Hospital, Shimoina Gun, Nagano Pref.
  - Yokoyama Medical Clinic, Shiojiri, Nagano Pref.
  - Sato Clinic, Suzaka, Nagano Pref.
  - Hoshiko Clinic, Nagasaki, Nagasaki Pref.
  - Shinagawa Clinic, Nagasaki, Nagasaki Pref.
  - Iryohojin Yamamoto Naika, Nishisonogi Gun, Nagasaki Pref.
  - Yamada Clinic, Gojō, Nara Pref.
  - Uyama Naika Clinic, Ikoma, Nara Pref.
  - Clinic Jinguumae, Kahihara City, Nara Pref.
  - Kasahara Clinic, Kahihara City, Nara Pref.
  - Sawada Clinic, Kashiba, Nara Pref.
  - Doi Clinic, Kashihara, Nara Pref.
  - Medical Corporation Kiriyama Clinic, Kashihara, Nara Pref.
  - Miyamoto Clinic, Kashihara, Nara Pref.
  - Oosumi Naika Iin, Kashihara, Nara Pref.
  - Kondo Clinic Mamigaoka Purified Center, Kitakatsuragi Gun, Nara Pref.
  - Matsuoka Clinic, Kitakatsuragi Gun, Nara Pref.
  - Nakahori Iin, Kitakatsuragi Gun, Nara Pref.
  - Seiwadai Clinic, Kitakatsuragi Gun, Nara Pref.
  - Saiseikai Nara Hospital, Nara, Nara Pref.
  - Takanohara Central Hospital, Nara, Nara Pref.
  - Takanohara Suzuran-naika, Nara, Nara Pref.
  - Ote Clinic of Internal Medicine, Sakurai, Nara Pref.
  - Sakaguchi Clinic, Sakurai, Nara Pref.
  - Kokuho Central Hospital, Shiki Gun, Nara Pref.
  - Makiura Naika, Yamatokōriyama, Nara Pref.
  - Matsuta Heart Clinic, Yamatokōriyama, Nara Pref.
  - Nakatani Clinic, Yamatotakada City, Nara Pref.
  - Sano Clinic, Murakami, Niigata Pref.
  - Kawaguchi Clinic, Nagaoka, Niigata Pref.
  - Maeda Medical Clinic, Niigata, Niigata Pref.
  - Watanabe NJ Clinic, Beppu, Oiat Pref.
  - Hirata Clinic, Ōita, Oiat Pref.
  - Ninomiya Clinic, Ōita, Oiat Pref.
  - Sumi Cardiology Clinic, Ōita, Oiat Pref.
  - Tokumaru Digestive Internal Medicine Clinic, Ōita, Oiat Pref.
  - Tsuzaki Clinic, Ōita, Oiat Pref.
  - Ishida Medical Clinic, Usa, Oiat Pref.
  - Hachiouji Naika Clinic, Kurashiki, Okayama Pref.
  - Inada Clinic, Kurashiki, Okayama Pref.
  - Hisamatsu Medical Clinic, Okayama, Okayama Pref.
  - Yuhara Naika Clinic, Okayama, Okayama Pref.
  - Hattori Clinic, Setouchi, Okayama Pref.
  - Nishimura Clinic, Fujiidera, Osaka Pref.
  - Ikeda Clinic, Higashiosaka, Osaka Pref.
  - Ogawa Clinic, Higashiosaka, Osaka Pref.
  - Taisei Clinic, Hirakata, Osaka Pref.
  - Ishiga Clinic, Ibaraki, Osaka Pref.
  - Masuda Clinic, Ibaraki, Osaka Pref.
  - Kanazawa Clinic, Izumi, Osaka Pref.
  - Misugi Clinic, Kaizuka, Osaka Pref.
  - Yoshida Clinic, Kaizuka, Osaka Pref.
  - Mori Iin, Kishiwada, Osaka Pref.
  - Medical Corporation Joukokai Teranishi-geka naika, Moriguchi, Osaka Pref.
  - Iryouhoujin Suisyoukai Murata Hospital, Osaka, Osaka Pref.
  - Izuoka Clinic, Osaka, Osaka Pref.
  - Keiju Hospital, Osaka, Osaka Pref.
  - Kondo Clinic, Osaka, Osaka Pref.
  - Kubota Clinic, Osaka, Osaka Pref.
  - Matsushita Medical Clinic, Osaka, Osaka Pref.
  - Nishizawa Clinic, Osaka, Osaka Pref.
  - Osaka General Medical Center, Osaka, Osaka Pref.
  - Senpuku Clinic, Osaka, Osaka Pref.
  - Tai Internal Medicin Clinic, Osaka, Osaka Pref.
  - Ueda Clinic, Osaka, Osaka Pref.
  - Ohta Iin, Sakai, Osaka Pref.
  - Ban Clinic, Suita, Osaka Pref.
  - Iryohojin Nogi Naika Iin, Suita, Osaka Pref.
  - Kobayashi Clinic, Suita, Osaka Pref.
  - Ichida Internal Clinic, Takaishi, Osaka Pref.
  - Yada Clinic, Takaishi, Osaka Pref.
  - Ryo Clinic, Takatsuki, Osaka Pref.
  - Matsuo Clinic, Yao, Osaka Pref.
  - Enomoto Clinic, Ageo, Saitama Pref.
  - Medimo Hanyu Clinic, Hanyū, Saitama Pref.
  - Hirose Hospital, Kawagoe, Saitama Pref.
  - Iryohojin Hogi Shinryojo, Kawaguchi, Saitama Pref.
  - Tokutake Iin, Kawaguchi, Saitama Pref.
  - Gamo Tenjinbashi Clinic, Koshigaya, Saitama Pref.
  - Matsumoto Clinic, Koshigaya, Saitama Pref.
  - Medical Corporation Shibuya Clinic, Kumagaya, Saitama Pref.
  - Akimoto Clinic, Saitama, Saitama Pref.
  - Iwatsuki-minami Hospital, Saitama, Saitama Pref.
  - Suzuhiro Clinic, Saitama, Saitama Pref.
  - Nashida naika clinic, Tokorozawa, Saitama Pref.
  - Shizuoka Medical Alliance Shirahama Chuou Clinic, Shimoda, Shizuoka Pref.
  - Akiyama Clinic, Shizuoka, Shizuoka Pref.
  - Aoshima Clinic, Shizuoka, Shizuoka Pref.
  - Eguchi Clinic, Shizuoka, Shizuoka Pref.
  - Shizuoka Hospital, Shizuoka, Shizuoka Pref.
  - Ueno Clinic, Yaizu, Shizuoka Pref.
  - Takahashi Medical Clinic, Ohtawara City, Tochigi Pref.
  - Iryouhoujin Yuukoukai Morioka Naika Shonika, Oyama, Tochigi Pref.
  - Takada Clinic, Tochigi, Tochigi Pref.
  - Masuda Naika, Utsunomiya, Tochigi Pref.
  - Murakami Clinic, Anan, Tokushima Pref.
  - Fukushima Clinic, Itano Gun, Tokushima Pref.
  - Yamamoto Naika Ityoka, Itano Gun, Tokushima Pref.
  - Yuki National Health Insurance Hospital Of Minami Town, Kaifu Gun, Tokushima Pref.
  - Sekishinkan Hospital, Komatsushima, Tokushima Pref.
  - Ueta Clinic, Myozai Gun, Tokushima Pref.
  - Kensei Uchimachi Clinic, Tokushima, Tokushima Pref.
  - Kitagawa Naika Ityoka, Tokushima, Tokushima Pref.
  - Kitasako Clinic, Tokushima, Tokushima Pref.
  - Limbs Tokushima Clinic, Tokushima, Tokushima Pref.
  - Matsumura Internal, Gastrointestial Medicine, Tokushima, Tokushima Pref.
  - Okagawa Clinic, Tokushima, Tokushima Pref.
  - Yokoi Internal Medicine, Tokushima, Tokushima Pref.
  - Kimura Internal Medicine Clinic, Yoshinokawa City, Tokushima Pref.
  - Yata Clinic, Yoshinokawa City, Tokushima Pref.
  - Okubo Clinic, Akishima, Tokyo
  - Juntendo University Hospital, Bunkyo Ku, Tokyo
  - Choei Clinic, Edogawa Ku, Tokyo
  - Shiraishi Iin, Edogawa Ku, Tokyo
  - Hattori Clinic, Hachiōji, Tokyo
  - Toyoizumi Hospital, Hachiōji, Tokyo
  - Utsugidai Tajima Clinic, Hachiōji, Tokyo
  - Mochizuki Naika Clinic, Itabashi Ku, Tokyo
  - Nishio Clinic, Itabashi Ku, Tokyo
  - Ono Heart Clinic, Koto Ku, Tokyo
  - Shiba Palace Clinic, Minato-ku, Tokyo
  - Kamada Clinic, Mitaka, Tokyo
  - Tenjinmae Clinic, Mitaka, Tokyo
  - Takayama Iin, Mitaka-shi, Tokyo
  - Sugawara Clinic, Nerima Ku, Tokyo
  - Yamada Clinic, Ōta-ku, Tokyo
  - Matsumura Gastroenterological Clinic, Setagaya Ku, Tokyo
  - Magari Clinic, Shinjuku Ku, Tokyo
  - Yotsuya Internal Medicine Clinic, Shinjuku Ku, Tokyo
  - Yotsuya-Murakami Internal Medicine Clinic, Shinjuku Ku, Tokyo
  - Obayashi Clinic, Sumida City, Tokyo
  - Sumidagawa Clinic, Sumida Ku, Tokyo
  - ISHII Medical Clinic, Tachikawa-shi, Tokyo
  - Takahashi Ko Minako Clinic, Murayama, Yamagata Pref.
  - Obanazawa City Clinic, Obanazawa, Yamagata Pref.
  - Okuyama Clinic, Obanazawa, Yamagata Pref.
  - Sakae Clinic, Obanazawa, Yamagata Pref.
  - Honma Clinic, Sakata, Yamagata Pref.
  - Isoda Clinic, Yamagata, Yamagata Pref.
  - Nihei Clinic, Yamagata, Yamagata Pref.
  - Shimasaki Clinic, Yamagata, Yamagata Pref.
  - Yamagata Tokushukai Hospital, Yamagata, Yamagata Pref.
  - Iwasaki Naika Iin, Iwakuni, Yamaguchi Pref.
  - Kuwahara Clinic, Iwakuni, Yamaguchi Pref.
  - Ayame Medical Clinic, Shimonoseki, Yamaguchi Pref.
  - Johno Clinic, Shimonoseki, Yamaguchi Pref.
  - Matsuda Medical Clinic, Shimonoseki, Yamaguchi Pref.
  - Mizumachi Medical Clinic, Shimonoseki, Yamaguchi Pref.
  - Noda Clinic, Shimonoseki, Yamaguchi Pref.
  - Fujii Clinic, Ube, Yamaguchi Pref.
  - Shakaiiryouhoujin Onaka Hospital, Ube, Yamaguchi Pref.
  - Watada-naika Hospital, Ube, Yamaguchi Pref.
  - Ouchi Clinic, Yamaguchi, Yamaguchi Pref.
  - Yoshizaki Clinic, Chūō, Yamanashi Pref.
  - Takahashi Clinic, Nishi Yatsushiro Gun, Yamanashi Pref.
  - Higashikatsura Medical Clinic, Tsuru, Yamanashi Pref.
  - Fukushi Clinic, Aomori
  - Kashiwagi Clinic, Ayase
  - Hayashi Diabetes Clinic, Chigasaki
  - Uchiyama Clinic, Jōetsu
  - Nitta Medical Clinic, Kamiinagun
  - Imai Clinic, Kawasaki
  - Tani Clinic, Kitakyushu
  - Marumo Clinic, Koganei
  - Ihara Clinic, Kyoto
  - Goko-Hospital, Matsudo
  - Satou Clinic, Mooka
  - Iino Clinic, Nirasaki
  - Miura Clinic, Osaka
  - Kuroda Iin, Ōtsuki
  - Sasaki Clinic, Sendai
  - Kamata Clinic of Internal Medicine, Shiki
  - Nishikawa Clinic, Shimoda
  - Satou Iin, Shimoinagun
  - Kumagai Clinic, Shinshiro
  - Suzuki Clinic, Toyokawa
  - Benibana Clinic, Yamagata
  - Fujimi Clinic, Yokohama
  - Hongo Clinic, Yokohama
  - Jiyukai Yamada Naika, Yokohama
  - Shonan Ochanomizu Clinic, Yokohama
  - Tani Clinic Internal Medicine, Allergology & Rheumatology, Yokohama